CLINICAL TRIAL: NCT06604936
Title: Investigation of Balance and Core Endurance in Patients With Fibromyalgia Syndrome
Brief Title: Investigation of Core Endurance in Fibromyalgia
Status: Recruiting | Type: Observational
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Head of Physiotherapy and Rehabilitation Department, Firat University
Other Study IDs: 2022/ 11- 24
Record Dates: First submitted 2024-08-14; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; core endurance test; balance
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia group: Demographic information (age, height, weight, occupation, medication, smoking) of the individuals who agreed to participate in the study will be recorded. Then, static and dynamic core endurance tests will be performed to evaluate core endurance. Static core endurance tests will include side bridge test, trunk flexion test, trunk extension test and prone bridge test. Modified push-ups and sit-ups tests will be performed as dynamic core endurance tests. Functional status of the patients will be evaluated with the Fibromyalgia Impact Questionnaire. Static and dynamic balance assessment will be evaluated using the HUR BTG4 Balance Master System and Berg Balance Scale.
  Interventions: Other: Fibromyalgia group
- Healthy group: individuals who agreed to participate in the study will be recorded. Then, static and dynamic core endurance tests will be performed to evaluate core endurance. Static core endurance tests will include side bridge test, trunk flexion test, trunk extension test and prone bridge test. Modified push-ups and sit-ups tests will be performed as dynamic core endurance tests. Static and dynamic balance assessment will be evaluated using the HUR BTG4 Balance Master System and Berg Balance Scale.
  Interventions: Other: Healthy group

INTERVENTIONS:
Other: Fibromyalgia group — Demographic information (age, height, weight, occupation, medication, smoking) of the individuals who agreed to participate in the study will be recorded. Then, static and dynamic core endurance tests will be performed to evaluate core endurance. Static core endurance tests will include side bridge test, trunk flexion test, trunk extension test and prone bridge test. Modified push-ups and sit-ups tests will be performed as dynamic core endurance tests. Functional status of the patients will be evaluated with the Fibromyalgia Impact Questionnaire. Static and dynamic balance assessment will be evaluated using the HUR BTG4 Balance Master System and Berg Balance Scale.
  Groups: Fibromyalgia group
Other: Healthy group — Demographic information (age, height, weight, occupation, medication, smoking) of the individuals who agreed to participate in the study will be recorded. Then, static and dynamic core endurance tests will be performed to evaluate core endurance. Static core endurance tests will include side bridge test, trunk flexion test, trunk extension test and prone bridge test. Modified push-ups and sit-ups tests will be performed as dynamic core endurance tests. Static and dynamic balance assessment will be evaluated using the HUR BTG4 Balance Master System and Berg Balance Scale.
  Groups: Healthy group

SUMMARY:
The aim of this study is to compare core endurance and balance in patients with Fibromyalgia Syndrome (FMS) with healthy subjects and to evaluate the relationship between core endurance and balance.The study will include 44 FMS patients and 44 age- and sex-matched healthy controls. Demographic data of the participants will be recorded. Then, core endurance will be assessed with McGill core endurance tests, balance will be evaluated with HUR BTG4 Balance Master System and Berg Balance Scale (BBS), and function will be assessed with Fibromyalgia Impact Questionnaire (FIQ).

DETAILED DESCRIPTION:
Fibromyalgia Syndrome (FMS) is defined as a chronic disease with an unclear etiology, which is characterized by widespread musculoskeletal pain, mainly non-inflammatory, in females between 40-60 years of age, accompanied by fatigue, weakness, sleep problems, depression, anxiety and various cognitive and somatic disorders. The etiology and pathophysiology are still unclear. Balance is a key component of activities of daily living such as walking, running and climbing stairs. Maintaining an upright posture is a complex process that involves perceiving and integrating sensory inputs, planning movements, and executing them effectively. It is also defined as the ability to control the center of gravity within the base of support. The aim of this study is to compare core endurance and balance in patients with Fibromyalgia Syndrome (FMS) with healthy subjects and to evaluate the relationship between core endurance and balance.The study will include 44 FMS patients and 44 age- and sex-matched healthy controls. Demographic data of the participants will be recorded. Then, core endurance will be assessed with McGill core endurance tests, balance will be evaluated with HUR BTG4 Balance Master System and Berg Balance Scale (BBS), and function will be assessed with Fibromyalgia Impact Questionnaire (FIQ).

ELIGIBILITY:
Inclusion Criteria:

* Patients who were aged between 18-65 years,
* Patients who got diagnosed with Fibromyalgia Syndrome

Exclusion Criteria:

* Patients who had regular exercise habits, malignancy, pregnancy, incorporation
* Patients who had changes of medical treatment in last 3 months
* Patients who had dysfunction that can prevent physical activity

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 years, diagnosed with FMS by clinical and physical examination, who agreed to participate in the study were included in the study. Patients with a diagnosis of severe spinal stenosis, concomitant systemic inflammatory rheumatic disease, pregnancy, malignancy or infection, history of surgery in the last 3 months, and physical problems that would prevent the application of core endurance tests were excluded.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-17 (Estimated); Primary Completion 2024-10-14 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Side bridge test | up to 2 weeks
  Participants will be asked to lift their hips off the floor in a side lying position with support from the elbow and forearm. After the patients will place their whole body in a straight line on their feet and elbows, the time was started to be kept with a stopwatch. The time will be maintained for the right and left side was recorded as a score.
Trunk flexion test | up to 2 weeks
  Participants will be asked to position the upper trunk at 60⁰ flexion while the hips and knees will be in the 90⁰ flexion position. The time the patients could stand while maintaining this angle will be recorded.
Trunk extension test | up to 2 weeks
  Participants will be asked to lie prone out of the bed from the upper part of the iliac crista with their hips and knees in full extension. The time will maintain the horizontal position with their arms in the inverted T position will be measured with a stopwatch and recorded

SECONDARY OUTCOMES:
Balance assessment | up to 2 weeks
  Balance will be evaluated with the HUR BTG4 Balance Master System® (HUR International, Finland) on stable and unstable platform.
Functional assessment | up to 2 weeks
  Function will be assessed with the Fibromyalgia Impact Questionnaire (FIQ). The FIQ consists of 10 items. The first item includes daily activity questions scored on a Likert scale from 0 to 3 (always able to do - never able to do). The 10 items are added together to calculate the total score
Demographic assessment | up to 2 weeks
  Age, height, weight, occupation, medication, smoking will be asked and recorded from the patients

CONTACTS AND LOCATIONS:
Locations (1):
- Songul Baglan Yentur, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No